CLINICAL TRIAL: NCT06661694
Title: A PHASE 1, RANDOMIZED, OPEN-LABEL, 4-PERIOD, CROSSOVER, SINGLE-DOSE STUDY IN HEALTHY PARTICIPANTS TO ESTIMATE THE EFFECT OF TABLET FORMULATION ON THE RELATIVE BIOAVAILABILITY OF MEVROMETOSTAT (PF-06821497)
Brief Title: A Study to Learn How Different Tablets of the Study Medicine Mevrometostat Are Taken up Into the Blood in Healthy Adults
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: sponsor decision
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: C2321006; 2024-516907-18-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2024-10-24; First posted 2024-10-28 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2024-11

CONDITIONS: Healthy
MeSH Terms: interventions — PF06821497

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sequence 1 (Experimental): Participants will receive a single 875 mg dose of Treatment A on Day 1 of Period 1, followed by a single 875 mg dose of Treatment B on Day 1 of Period 2, followed by a single 875 mg dose of Treatment C on Day 1 of Period 3, followed by a single 875 mg dose of Treatment D on Day 1 of Period 4.
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C; Drug: Treatment D
- Sequence 2 (Experimental): Participants will receive a single 875 mg dose of Treatment B on Day 1 of Period 1, followed by a single 875 mg dose of Treatment D on Day 1 of Period 2, followed by a single 875 mg dose of Treatment A on Day 1 of Period 3, followed by a single 875 mg dose of Treatment C on Day 1 of Period 4.
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C; Drug: Treatment D
- Sequence 3 (Experimental): Participants will receive a single 875 mg dose of Treatment C on Day 1 of Period 1, followed by a single 875 mg dose of Treatment A on Day 1 of Period 2, followed by a single 875 mg dose of Treatment D on Day 1 of Period 3, followed by a single 875 mg dose of Treatment B on Day 1 of Period 4.
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C; Drug: Treatment D
- Sequence 4 (Experimental): Participants will receive a single 875 mg dose of Treatment D on Day 1 of Period 1, followed by a single 875 mg dose of Treatment C on Day 1 of Period 2, followed by a single 875 mg dose of Treatment B on Day 1 of Period 3, followed by a single 875 mg dose of Treatment A on Day 1 of Period 4.
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C; Drug: Treatment D

INTERVENTIONS:
Drug: Treatment A — Single 875 mg dose of mevrometostat standard tablet formulation
  Other Names: PF-06821497
Drug: Treatment B — Single 875 mg dose of mevrometostat alternative tablet formulation
  Other Names: PF-06821497
Drug: Treatment C — Single 875 mg dose of mevrometostat alternative tablet formulation
  Other Names: PF-06821497
Drug: Treatment D — Single 875 mg dose of mevrometostat alternative tablet formulation
  Other Names: PF-06821497

SUMMARY:
The purpose of the study is to compare the amount of mevrometostat available from four different tablet formulations, taken with food, in healthy adult participants.

This study is seeking male or female participants who:

* are 18 years or older
* are healthy as decided by medical tests.
* have a Body mass index (BMI) of 16 to 32 kilogram per meter squared
* a total body weight of more than 50 kilograms (110 pounds).

All participants will take part in 4 study periods to receive 4 different treatments, which are assigned in a random order. There will also be a 5-day gap between each study period. This is done so that the medicine is passed out of the body before the start of the next period.

Each treatment consists of a single dose of mevrometostat (PF-06821497), and the treatments differ only by tablet formulation.

How the medicine is processed in the body will be studied after giving the medicines to the participants. This will be done by collecting blood samples after giving each of these tablets. The results will be used to see the effect of tablet formulation on the amount of mevrometostat (PF-06821497) available in the blood of the participants.

Participants will be in the study for about 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participants ≥18 years of age, inclusive, at screening.
* Male and female participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, vital signs and 12-lead ECGs.
* BMI of 16-32 kg/m2; and a total body weight >50 kg (110 lb)
* Evidence of a personally signed and dated ICD indicating that the participant has been informed of all pertinent aspects of the study.
* Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing) or prior allergic reaction to any component of mevrometostat.

  * Any condition possibly affecting drug absorption (eg, gastrectomy, cholecystectomy).
  * History of HIV infection, hepatitis B, or hepatitis C; positive testing for HIV, HBsAg, HBsAb, HBcAb, or HCVAb. Hepatitis B vaccination is allowed.
* Any medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality or other conditions that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* Previous administration with an investigational product (drug or vaccine) within 30 days (or as determined by the local requirement) or 5 halflives preceding the first dose of study intervention used in this study (whichever is longer). Participation in studies of other investigational products (drug or vaccine) at any time during participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-04-28 (Estimated); Primary Completion 2025-09-08 (Estimated); Study Completion 2025-09-09 (Estimated)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Mevrometostat (Formulation 1) | Period 1-4: pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, and 72 hour(s) post-dose
  To estimate the bioavailability of a single 875 mg dose of mevrometostat (Formulation 2) relative to a single 875 mg dose of mevrometostat (Formulation 1) under fed conditions in healthy adult participants.
Maximum Observed Plasma Concentration (Cmax) of Mevrometostat (Formulation 2) | Period 1-4: pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, and 72 hour(s) post-dose
  To estimate the bioavailability of a single 875 mg dose of mevrometostat (Formulation 2) relative to a single 875 mg dose of mevrometostat (Formulation 1) under fed conditions in healthy adult participants.
Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) of Mevrometostat (Formulation 1) | Period 1-4: pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, and 72 hour(s) post-dose
  To estimate the bioavailability of a single 875 mg dose of mevrometostat (Formulation 2) relative to a single 875 mg dose of mevrometostat (Formulation 1) under fed conditions in healthy adult participants.
Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) of Mevrometostat (Formulation 2) | Period 1-4: pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, and 72 hour(s) post-dose
  To estimate the bioavailability of a single 875 mg dose of mevrometostat (Formulation 2) relative to a single 875 mg dose of mevrometostat (Formulation 1) under fed conditions in healthy adult participants.

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Mevrometostat (Formulation 3) | Period 1-4: pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, and 72 hour(s) post-dose
  To estimate the bioavailability of a single 875 mg dose of mevrometostat (Formulation 3) relative to a single 875 mg dose of mevrometostat (Formulation 2) and to estimate the bioavailability of a single 875 mg dose of mevrometostat (Formulation 4) relative to a single 875 mg dose of mevrometostat (Formulation 2) under fed conditions in healthy adult participants.
Maximum Observed Plasma Concentration (Cmax) of Mevrometostat (Formulation 4) | Period 1-4: pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, and 72 hour(s) post-dose
  To estimate the bioavailability of a single 875 mg dose of mevrometostat (Formulation 3) relative to a single 875 mg dose of mevrometostat (Formulation 2) and to estimate the bioavailability of a single 875 mg dose of mevrometostat (Formulation 4) relative to a single 875 mg dose of mevrometostat (Formulation 2) under fed conditions in healthy adult participants.
Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) of Mevrometostat (Formulation 3) | Period 1-4: pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, and 72 hour(s) post-dose
  To estimate the bioavailability of a single 875 mg dose of mevrometostat (Formulation 3) relative to a single 875 mg dose of mevrometostat (Formulation 2) and to estimate the bioavailability of a single 875 mg dose of mevrometostat (Formulation 4) relative to a single 875 mg dose of mevrometostat (Formulation 2) under fed conditions in healthy adult participants.
Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) of Mevrometostat (Formulation 4) | Period 1-4: pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, and 72 hour(s) post-dose
  To estimate the bioavailability of a single 875 mg dose of mevrometostat (Formulation 3) relative to a single 875 mg dose of mevrometostat (Formulation 2) and to estimate the bioavailability of a single 875 mg dose of mevrometostat (Formulation 4) relative to a single 875 mg dose of mevrometostat (Formulation 2) under fed conditions in healthy adult participants.
Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs) | Time the participant provides informed consent through and including follow-up contact occurring 28-35 calendar days after the lasts administration of the study intervention.
  To evaluate the safety and tolerability of mevrometostat when administered as a tablet formulation to healthy participants.
Number of Participants With Clinical Laboratory Abnormalities | Time the participant provides informed consent through and including follow-up contact occurring 28-35 calendar days after the lasts administration of the study intervention.
  To evaluate the safety and tolerability of mevrometostat when administered as a tablet formulation to healthy participants.
Number of Participants With Clinically Significant Change From Baseline in Vital Signs | Time the participant provides informed consent through and including follow-up contact occurring 28-35 calendar days after the lasts administration of the study intervention.
  To evaluate the safety and tolerability of mevrometostat when administered as a tablet formulation to healthy participants.
Number of Participants With Electrocardiogram (ECG) Abnormalities | Time the participant provides informed consent through and including follow-up contact occurring 28-35 calendar days after the lasts administration of the study intervention.
  To evaluate the safety and tolerability of mevrometostat when administered as a tablet formulation to healthy participants.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit - Brussels, Brussels, Bruxelles-capitale, Région de, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C2321006